CLINICAL TRIAL: NCT01093508
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Study to Assess the Tolerability and Pharmacokinetics of APD916 Administered to Healthy Adult Subjects
Brief Title: Single-dose Safety Study of APD916 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Ronald Shazer, MD, Arena Pharmaceuticals, Inc.
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD916-001
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Narcolepsy With or Without Cataplexy
MeSH Terms: interventions — (R)-1-(2-(4'-(3-methoxypropylsulfonyl)biphenyl-4-yl)ethyl)-2-methylpyrrolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: APD916

SUMMARY:
The APD916-001 study is designed primarily to evaluate the safety and tolerability of APD916 when administered as a single dose

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-dose escalation study of up to 9 dose cohorts (1, 2, 5, 10, 20, 30, 45, 70 and 90 mg) each comprising 8 subjects (2 to receive placebo, 6 to receive APD916). Each cohort will be assigned to receive a single dose of APD916. After dosing within the first cohort has been completed and safety data review identifies no tolerability issues, and the principal investigator (PI) and Sponsor have agreed that it is safe to proceed, then subjects in the next cohort may be dosed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females ages 18-45 years
* Body weight of 50-100 kg (110-220 pounds)
* Eligible female subjects will be non-pregnant, evidenced by a negative serum pregnancy test at Screening and a urine dipstick pregnancy test on Day -1 (Check-In); non-lactating; surgically sterile, postmenopausal, or agree to continue to use a medically accepted method of birth control during and for at least 1 month after last study medication administration.
* Eligible male subjects will either be surgically sterile (i.e., vasectomy), for at least 3 months prior to screening, or agree to use a condom with spermicide when sexually active with a female partner who is not using an acceptable method of birth control during the study and for 1 month after.

Exclusion Criteria

* Subject who has donated any blood, or had significant blood loss within 56 days of dosing
* History of smoking or tobacco use within 3 months prior to dosing
* History of epilepsy or other seizure disorder
* Recent history (within 2 years prior to the screening visit) of sleep disorders
* History (within 2 years prior to the screening visit) of ADD or ADHD
* Traveled across more than 3 time zones within 2 weeks prior to dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single, escalating doses of APD916 when administered to healthy adult subjects | Single dose
  Safety measures to include adverse events, vital signs, 12-lead ECGs, physical examinations, and clinical lab parameters.

SECONDARY OUTCOMES:
To assess the pharmacokinetic properties of single, escalating doses of APD916 | Single dose
  Pharmacokinetic samples (blood and urine) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: James Maynard, MD, Principal Investigator — Community Research, Cincinnati, OH
Locations (1):
- Community Research, Cincinnati, Ohio, United States

REFERENCES:
- See also: Related Info — http://www.arenapharm.com